CLINICAL TRIAL: NCT07130526
Title: Trial to Investigate the Shockwave Intravascular Lithotripsy (IVL) on Vascular Compliance in Heavily Calcified Femoropopliteal Disease (PACSS 2-4)
Brief Title: Distrupt Stiffness Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Collaborators: Shockwave Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FRM-68717
Record Dates: First submitted 2025-06-04; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: PAD - Peripheral Arterial Disease; PAD
Keywords: pad; peripheral artery disease; intravascular lithotripsy
MeSH Terms: conditions — Peripheral Vascular Diseases; Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POBA plus DCB (Active Comparator)
  Interventions: Device: POBA plus DCB
- Intravascular Lithotripsy (IVL) plus DCB (Active Comparator)
  Interventions: Device: Intravascular Lithotripsy (IVL) plus DCB

INTERVENTIONS:
Device: Intravascular Lithotripsy (IVL) plus DCB — The device under investigation is the Peripheral Lithotripsy System (Shockwave Medical, Fremont, California). Miniaturized and arrayed lithotripsy emitters create a localized field effect at the site of the calcium. The Peripheral Lithotripsy System is CE-marked for peripheral arterial disease and for this study, will be used within its indication for use. This included the following: intended for lithotripsy-enhanced balloon dilatation of lesions, including calcified lesions, in the peripheral vasculature, including the iliac, femoral, ilio-femoral and popliteal arteries.
  The IVL catheter is delivered across a calcified lesion over an 0.014'' wire and the integrated balloon is expanded to 4atm to facilitate efficient energy transfer.
  An electrical discharge from the emitters vaporizes the fluid within the balloon, creating a rapidly expanding and collapsing bubble that generates sonic pressure waves. The waves create a localized field effect that travels through soft vascular tissue,
  Arms: Intravascular Lithotripsy (IVL) plus DCB
Device: POBA plus DCB — Standard of Care
  Arms: POBA plus DCB

SUMMARY:
Typical symptoms of PAD include exercise-induced pain in the legs (known as intermittent claudication), which can significantly limit pain-free walking. In more advanced stages, pain may also occur at rest. Additionally, the development of chronic, hard-to-heal wounds-especially on the feet and toes-is possible. These wound healing impairments are caused by the insufficient supply of oxygen and nutrients to the affected tissues.

The underlying cause of PAD is usually atherosclerosis, a pathological change in the vessel walls due to the accumulation of fats, calcium, and connective tissue. These deposits lead to stiffening and narrowing of the arteries, severely restricting blood flow. Major risk factors for the development of PAD include widespread chronic conditions such as diabetes mellitus, hyperlipidemia (elevated blood lipid levels, e.g., cholesterol), arterial hypertension (high blood pressure), obesity, and tobacco use.

Various therapeutic options are available for the treatment of PAD. In addition to conservative therapy (such as supervised exercise training, pharmacological blood thinning, and risk factor management), interventional, minimally invasive treatment using catheter-based techniques is frequently employed. In such procedures, a thin catheter is guided through the vascular system to the affected area of the leg artery. Depending on the type and extent of the arterial narrowing or calcification, one of the following techniques may be applied:

Balloon angioplasty: Dilation of the vessel using an inflatable balloon. Lithoplasty: Application of shockwaves to break down calcifications in the arterial wall.

DETAILED DESCRIPTION:
Massive Calcifications in the peripheral vessels lead to altered vascular stiffness. This arterial stiffness is an excellent marker for morbidity and mortality and correlates with the progression of cardiovascular disease. Main pathophysiologic principles are altered pulse wave reflections through arterial and aortic stiffness on cardiac functions. Impaired vascular compliance is associated with increased cardiovascular morbidity and leads to a progression of atherosclerotic lesions, impaired ventriculoarterial coupling and ultimately impaired coronary perfusion.

Vascular calcifications are furthermore held responsible for suboptimal vessel expansion and increased risk of complications including dissection and perforation and reduced long-term patency when treated though the endovascular route. Calcium treatment through IVL gives physicians opportunities to tackle this unmet need. IVL treatment is a safe and effective treatment in these heavily calcified lesions proving excellent procedural success compared to PTA driven by a significantly lower rate of major dissections and need for bail-out stent placement. This was evident also in coronary vessels suggesting that calcium fracture is the IVL-related mechanism to enhance vessel compliance and to assists optimal stent expansion.

The influence of this novel strategies with improved hemodynamic capabilities with respect to vasomotion of the vessel wall, vascular function and vascular compliance can be measured by ultrasound, as shown recently. To which extent intravascular lithotripsy has an impact on vessel compliance has not been elucidated so far and could aid to understand the prognostic beneficial effects of intravascular lithotripsy.

The aim of this investigator-initiated trial is thus to investigate the IVL -related beneficial effect of lesion preparation by altering vascular compliance parameters and vasomotion of the vessel wall.

The primary objective is to determine changes in Vessel compliance, function and stiffness and after IVL treatment compared to POBA in symptomatic PAD.

Local vascular compliance as determined through FDC (fractional diameter change) in the distal IEA, CFA, prox. SFA or PA. Measurement of vascular compliance or function in patients is a powerful tool for atherosclerosis research. FDC represents the ratio of the vessel's diameter change between systole and diastole divided by the diastolic diameter. Several interventions are known to decrease cardiovascular risk, including exercise, smoking cessation, or medications with statins improving vascular compliance. Therefore, vascular compliance serves as a ''barometer'' for cardiovascular health that can be used for evaluation of new therapeutic strategies and is prognostic relevant. Moreover numerous studies have proven the prognostic value of vasomotor dysfunction, demonstrating that impaired vasomotor function identifies patients who have increased risk for cardiovascular events. Until now, it is completely unknown if intravascular lithotripsy has an impact on local vascular functions. We have recently shown an impact of paclitaxel coated ballons and mechanical atherothrombectomy on local vascular functions.

Further outcome measures include local and systemic vascular function and stiffness determined through pulse wave velocity (PWV), flow-mediated dilatation (FMD) and augmentation index (augmentation index). Vascular and aortic stiffness, assessed by measurement of PWV, can predict future cardiovascular events and mortality, even after accounting for other established cardiovascular risk factors. During the last years, a large amount of evidence has accumulated demonstrating that arterial stiffness is an important risk factor for cardiovascular disease. FMD represents the percent diameter gain as calculated based on pre-ischemia and post-ischemia (and reactive hyperemia) diameter measurements of the femoral artery. In this context, ischemia is induced through vessel occlusion by means of inflating a blood pressure cuff around the forearm or leg. Standard techniques as determined by Doppler and duplex ultrasonography will quantify tissue perfusion and primary patency. Furthermore, technical success, procedural complications and freedom from target lesion revascularization will be determined.

Peripheral Lithotripsy System The device under investigation is the Peripheral Lithotripsy System (Shockwave Medical, Fremont, California). Miniaturized and arrayed lithotripsy emitters create a localized field effect at the site of the calcium. The Peripheral Lithotripsy System is CE-marked for peripheral arterial disease and for this study, will be used within its indication for use. This included the following: intended for lithotripsy-enhanced balloon dilatation of lesions, including calcified lesions, in the peripheral vasculature, including the iliac, femoral, ilio-femoral and popliteal arteries.

The IVL catheter is delivered across a calcified lesion over an 0.014'' wire and the integrated balloon is expanded to 4atm to facilitate efficient energy transfer.

An electrical discharge from the emitters vaporizes the fluid within the balloon, creating a rapidly expanding and collapsing bubble that generates sonic pressure waves. The waves create a localized field effect that travels through soft vascular tissue, selectively cracking intimal and medial calcium within the vessel wall.

After calcium modification, the integrated balloon may subsequently be used to dilate the lesion at low pressure to maximize luminal gain.

ELIGIBILITY:
Inclusion Criteria:

* Peripheral artery disease
* Severe Calcification PACCS 2,3 and 4
* Target lesions in distal EIA, CFA, prox. SFA or PA
* Clinical diagnosis of chronic, symptomatic lower limb ischemia as defined by Rutherford 2, 3, 4 and 5
* Planed peripheral intervention TASC A-D
* Subject must be between 18 and 85 years old
* Willing to comply with the specified follow-up evaluation
* Written informed consent prior to any study procedures

Exclusion Criteria:

* Target lesions with no optimal visualization in ultrasound
* Instent-Restenosis
* Thrombolysis within 72 hours prior to the index procedure
* Aneurysm formations in the femoral artery or popliteal artery
* Concomitant hepatic insufficiency, deep venous thrombus, coagulation disorder or receiving immunosuppressant therapy
* Unstable angina pectoris at the time of the enrolment
* Recent myocardial infarction or stroke < 30 days prior to the index procedure
* Life expectancy less than 12 months
* Septicemia at the time of enrolment
* Known or suspected active infection at the time of the index procedure, excluding an infection of a lower extremity wound of the target limb
* Known or suspected allergies or contraindications to aspirin, clopidogrel or heparin

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
FDC | 1 day and 30 days follow-up
  To determine changes in vessel compliance before and after IVL treatment and after 1 month compared to POBA in symptomatic PAD as determined by fractional diameter change (FDC).

SECONDARY OUTCOMES:
FMD/NMD analysis of the target lesion | 1 day and 30 days follow-up
  • Endothelial function and endothelial independent function as determined by FMD/NMD analysis of the target lesion. FMD represents the percent diameter gain as calculated based on preischemia and postischemia diameter measurements of the femoral artery. NMD represents the diameter change of the femoral artery after nitroglycerine-mediated vasodilation.
PWV | 1 day and 30 days follow-up
  Aortic stiffness determined by pulse wave velocity (PWV)
ABI | 1 day and 30 days follow-up
  Peripheral perfusion determined by ABI (ankle brachial index)
Primary patency (PP) | 1 day and 30 days follow-up
  Primary patency (PP) evaluated by clinical assessment by ultrasound
AIX | 1 day and 30 days follow-up
  Arterial stiffness determined by augmentation index (AIX@75HR). Changes in cardiovascular function measured by augmentation index in percent
Procedural complications | 1 day and 30 days follow-up
  Procedural complications
Dissection rate and Bail-out stenting | 1 day and 30 days follow-up
  Dissection rate and Bail-out stenting in % of treated patients
Freedom from Target Lesion Revascularization (FTLR) | 1 day and 30 days follow-up
  Freedom from Target Lesion Revascularization (FTLR)

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - West German Heart and Vascular Center, Clinic for Cardiology and Vascular Medicine, Universtiy Hospital Essen, Essen, North Rhine-Westphalia
  - University of Duisburg-Essen, Essen

IPD SHARING:
Plan to Share IPD: No